CLINICAL TRIAL: NCT06844591
Title: Comparison Between Conditioning Exercises and Resistance Interval Training on Quality of Life, Cardiorespiratory Fitness and Endurance in Post-CABG Patients
Brief Title: Effects of Conditioning Exercises and Resistance Interval Training on Post CABG Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0322 Rubab
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Bypass Grafting; Conditioning Therapy; Quality of Life; Resistance Training.
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Participants will complete a well-tested Performa. Basic parameters will be collected through the outcome measure tool. Group A will be given a Conditioning exercise protocol while the other Group B will be given resistance interval training for 6 weeks. The difference in improvement before and after 6 weeks will be documented and compared.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conditioning Exercise Group (Experimental): Aerobic interval training (AIT), which included rest intervals in between sessions of aerobic activity on a stationary bike and treadmill, was administered to the control group. A 10-minute warm-up, or a maximum of 50% to 60% of HR, preceded the program. Participants will complete a well-tested Performa. Basic parameters will be collected through the outcome measure tool. The difference in improvement before and after 6 weeks will be documented and compared.
  Interventions: Other: Conditioning Exercises/ Aerobic Interval Training
- Resistance Interval Training Group (Experimental): Resistance interval training for post-coronary artery bypass grafting (CABG) patients requires careful consideration and should be conducted under the supervision of healthcare professionals, such as cardiac rehabilitation specialists or physiotherapists. Exercise programs for individuals recovering from cardiac surgery must be tailored to their specific needs, taking into account their overall health, medical history, and current fitness level. Before beginning any exercise program, it's essential to obtain clearance from a healthcare provider. The workout lasted thirty to forty minutes in total. To fit the training load, resistance and intensity were gradually raised. For six weeks, this supervised training program was adhered to three times a week on alternate days. The difference in improvement before and after 6 weeks will be documented and compared.
  Interventions: Other: Resistance Interval Training

INTERVENTIONS:
Other: Conditioning Exercises/ Aerobic Interval Training — Aerobic interval training (AIT), which included rest intervals in between sessions of aerobic activity on a stationary bike and treadmill, was administered to the control group. A 10-minute warm-up, or a maximum of 50% to 60% of HR, preceded the program. The next activity round consisted of six x six-minute intervals of cycling and walking/uphill running on a treadmill at 60% to 85% of THR, separated by three minutes of rest/recovery. A ten-to fifteen-minute cool- down period followed the session.
  Arms: Conditioning Exercise Group
Other: Resistance Interval Training — Resistance interval training for post-coronary artery bypass grafting (CABG) patients requires careful consideration and should be conducted under the supervision of healthcare professionals, such as cardiac rehabilitation specialists or physiotherapists. Exercise programs for individuals recovering from cardiac surgery must be tailored to their specific needs, taking into account their overall health, medical history, and current fitness level. Before beginning any exercise program, it's essential to obtain clearance from a healthcare provider. The workout lasted thirty to forty minutes in total. To fit the training load, resistance and intensity were gradually raised. For six weeks, this supervised training program was adhered to three times a week on alternate days
  Arms: Resistance Interval Training Group

SUMMARY:
Coronary artery disease (CAD) is a global health challenge influenced by diabetes, hypertension, and psychosocial stress, with women having a higher prevalence of Coronary microvascular disease. Promoting coronary collateral circulation offers an alternative coronary artery disease CAD treatment. Invasive interventions like PCI and CABG aim to enhance coronary flow, restoring blood flow to ischemic myocardium. Post-CABG challenges include depression, anxiety, and factors affecting quality of life. Physiotherapy impacts heart rate variability, with virtual reality physiotherapy reducing both heart rate variability and hospital stay. Cardiac rehabilitation involves lifestyle changes, enhancing functional capacity, and supporting early recovery. Pre-operative respiratory muscle training improves outcomes. Acute high-intensity interval exercise and mild continuous exercise benefit exercise recovery. This research compares conditioning exercises and resistance interval training effects on post-CABG patients' well-being.

DETAILED DESCRIPTION:
The randomized clinical trial will be conducted in physical therapy department at the District Headquarters (DHQ) in Gujranwala, employing a non-probability convenience sampling technique. The study aims to include individuals aged 40-55 years. Participants in phase IV cardiac rehabilitation. Both female and male will be included.Exclusion criteria involve individuals with another clinical trial involving physical protocols. Regular practice of physical exercise of more than 150min per week in last 3 months. Decompensated heart failure. Further exclusions encompass individuals who have had an acute myocardial infarction or cardiac surgery within the last 6 months, severe valvular heart diseases, uncontrolled cardiac arrhythmias, asymmetric septal hypertrophic cardiomyopathy with dynamic obstruction in the outflow pathway, musculoskeletal disorders limiting completion of the exercise program, and impaired cognitive status affecting understanding and adherence to the study protocol. Group A will be given a Conditioning exercise protocol while the other Group B will be given resistance interval training. The difference in improvement before and after 6 weeks will be documented and compared.

ELIGIBILITY:
Inclusion Criteria:

* age 40-55 years
* post-coronary artery bypass graft (CABG) patients both females and males were included
* New York Heart Association criteria IV
* Hemodynamically stable patient

Exclusion Criteria:

* Fall in New York Heart Association criteria II III;
* Hemoglobin < 9 g/dL;
* Patients with peripheral or vascular problems of the lower limb,
* Cognitive and/or mental disorders;
* Exercise limiting comorbidities (primarily orthopedic, neurological condition)
* Enrollment in another clinical trial involving physical training protocols.
* Not willing to participate

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-09 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
SF-36 Questionnaire | 6 weeks
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used for quality of life, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study for the objective measure of the quality of life. The 36-Item Short Form Survey (SF-36) will be used which is a self-reported measure of health that covers eight domains of health.
6-minute walk test | 6 weeks
  The 6-minute walk test (6MWT) will be used for cardiorespiratory fitness, to measure the distance walked in a specified time and reflect the functional exercise level. The primary measurement is 6-min walk distance (6MWD), but during the 6MWT data can also be collected about the patient's blood oxygen saturation and perception of dyspnea during exertion. When conducting the 6MWT do not walk with the patient and do not assist the patient in carrying or pulling his or her supplemental oxygen. The patient should walk alone, not with other patients. Do not use a treadmill on which the patient adjusts the speed and/or the slope. Do not use an oval or circular track. An increase in the distance walked indicates improvement in basic mobility. Post training a difference of at least 45m should be observed for the 6 minutes' walk test to be sure that a "real" change in the patient's condition
30-second stand chair | 6 Weeks
  For endurance, the sit-to-stand (STS) test measures the number of times a person can stand up from a chair in a given time (30 seconds, 1 minute, or 5 repetitions). The 30 Second Sit to Stand Test is also known as 30 Second Chair Stand Test (30CST), was initially designed for testing leg strength and endurance in adults. The score is the total number of stands within 30 seconds (more than halfway up at the end of 30 seconds counts as a full stand).The 30-second chair stand involves recording the number of stands a person can complete in 30 seconds rather then the amount of time it takes to complete a pre- determined number of repetitions.

CONTACTS AND LOCATIONS:
Overall Officials: Qurat ul Ain, Principal Investigator — Riphah International University
Locations (1):
- Cheema Heart complex, Hospital Gujranwala, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terada T, Cotie L, Noda T, Vidal-Almela S, O'Neill CD, Reed JL. Effects of High-Intensity Interval Training, Moderate-to-Vigorous Intensity Continuous Training, and Nordic Walking on Functional Fitness in Patients with Coronary Artery Disease. J Cardiopulm Rehabil Prev. 2023 May 1;43(3):224-226. doi: 10.1097/HCR.0000000000000775. Epub 2023 Mar 2. No abstract available. PMID 36857093
- [Background] Kambic T, Bozic Mijovski M, Jug B, Hadzic V, Lainscak M. Anabolic and Inflammatory Response to High- and Low-Load Resistance Training in Patients with Coronary Artery Disease: A Randomized Controlled Trial. J Cardiopulm Rehabil Prev. 2023 Jul 1;43(4):307-309. doi: 10.1097/HCR.0000000000000783. Epub 2023 Mar 6. No abstract available. PMID 36867715
- [Background] McGregor G, Powell R, Begg B, Birkett ST, Nichols S, Ennis S, McGuire S, Prosser J, Fiassam O, Hee SW, Hamborg T, Banerjee P, Hartfiel N, Charles JM, Edwards RT, Drane A, Ali D, Osman F, He H, Lachlan T, Haykowsky MJ, Ingle L, Shave R. High-intensity interval training in cardiac rehabilitation: a multi-centre randomized controlled trial. Eur J Prev Cardiol. 2023 Jul 12;30(9):745-755. doi: 10.1093/eurjpc/zwad039. PMID 36753063
- [Background] Rengo JL, Savage PD, Hirashima F, Leavitt BJ, Ades PA, Toth MJ. Assessment of the Early Disabling Effects of Coronary Artery Bypass Graft Surgery Using Direct Measures of Physical Function. J Cardiopulm Rehabil Prev. 2022 Jan 1;42(1):28-33. doi: 10.1097/HCR.0000000000000587. PMID 33797459
- [Background] Kristiansen J, Sjuretharson T, Grove EL, Rasmussen J, Kristensen SD, Hvas AM, Mohr M. Feasibility and impact of whole-body high-intensity interval training in patients with stable coronary artery disease: a randomised controlled trial. Sci Rep. 2022 Oct 14;12(1):17295. doi: 10.1038/s41598-022-21655-w. PMID 36241898